CLINICAL TRIAL: NCT04294108
Title: Why Are Patients Still in Hospital After Video-Assisted Thoracoscopic Surgery Lobectomy?
Brief Title: Why in Hospital After VATS Lobectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lin Huang, Medical Doctor/ Research Fellow, Rigshospitalet, Denmark
Other Study IDs: H-20014489
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Pain, Postoperative; Postoperative Nausea and Vomiting; Infection; Air Leakage; Atrial Fibrillation
Keywords: in hospital; lobectomy; video-assisted thoracoscopic surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pain, Postoperative; Postoperative Nausea and Vomiting; Infections; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent VATS lobectomy: All consecutive patients scheduled for video-assisted thoracoscopic surgery lobectomy.
  Interventions: Other: Prolong in-hospital stay

INTERVENTIONS:
Other: Prolong in-hospital stay — Patients have a longer length of hospital stay than the common recommendation.

SUMMARY:
The study aims to identify specific or potential reasons that prolong the length of hospital stay after video-assisted thoracoscopic surgery lobectomy.

The hypothesis is that patients who are still in hospital after video-assisted thoracoscopic surgery lobectomy are associated with prolonged air leak, infection, pneumonia, atrial fibrillation or other complications or social factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to elective VATS lobectomy
* Speaks and understands Danish
* Informed consent obtained

Exclusion Criteria:

•Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent VATS lobectomy and writing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | Through study completion, an average of 2 days

SECONDARY OUTCOMES:
Number and frequency of postoperative complications | Up to 30 days
Numeric rating scale for postoperative pain in hospitalization | Through study completion, an average of 2 days
  Patients are scored using a numeric rating scale ranging from 0 (no pain) to 10 (excruciating pain) per day.
Drainage duration | Duration from postoperative chest tube placement to potential removal, an average of 2 days
  The criteria of drain removal is that air leak was consistently below 20 ml/min for at least 12 hours and fluid production was non-bloody and non-chylous without an upper volume limit.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Huang, MD, Principal Investigator — Rigshospitalet, Denmark; Henrik Kehlet, MD, DMSc, Study Director — Rigshospitalet, Denmark; Rene H Petersen, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laursen LO, Petersen RH, Hansen HJ, Jensen TK, Ravn J, Konge L. Video-assisted thoracoscopic surgery lobectomy for lung cancer is associated with a lower 30-day morbidity compared with lobectomy by thoracotomy. Eur J Cardiothorac Surg. 2016 Mar;49(3):870-5. doi: 10.1093/ejcts/ezv205. Epub 2015 Jun 18. PMID 26088592
- [Background] Agostini PJ, Lugg ST, Adams K, Smith T, Kalkat MS, Rajesh PB, Steyn RS, Naidu B, Rushton A, Bishay E. Risk factors and short-term outcomes of postoperative pulmonary complications after VATS lobectomy. J Cardiothorac Surg. 2018 Apr 12;13(1):28. doi: 10.1186/s13019-018-0717-6. PMID 29673386
- [Background] Kehlet H. ERAS Implementation-Time To Move Forward. Ann Surg. 2018 Jun;267(6):998-999. doi: 10.1097/SLA.0000000000002720. No abstract available. PMID 29462010
- [Background] Das-Neves-Pereira JC, Bagan P, Coimbra-Israel AP, Grimaillof-Junior A, Cesar-Lopez G, Milanez-de-Campos JR, Riquet M, Biscegli-Jatene F. Fast-track rehabilitation for lung cancer lobectomy: a five-year experience. Eur J Cardiothorac Surg. 2009 Aug;36(2):383-91; discussion 391-2. doi: 10.1016/j.ejcts.2009.02.020. Epub 2009 Mar 26. PMID 19324571
- [Background] Holbek BL, Horsleben Petersen R, Kehlet H, Hansen HJ. Fast-track video-assisted thoracoscopic surgery: future challenges. Scand Cardiovasc J. 2016;50(2):78-82. doi: 10.3109/14017431.2015.1114665. Epub 2015 Dec 1. PMID 26514281
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Husted H, Lunn TH, Troelsen A, Gaarn-Larsen L, Kristensen BB, Kehlet H. Why still in hospital after fast-track hip and knee arthroplasty? Acta Orthop. 2011 Dec;82(6):679-84. doi: 10.3109/17453674.2011.636682. Epub 2011 Nov 9. PMID 22066560
- [Background] Munk-Madsen P, Eriksen JR, Kehlet H, Gogenur I. Why still in hospital after laparoscopic colorectal surgery within an enhanced recovery programme? Colorectal Dis. 2019 Dec;21(12):1438-1444. doi: 10.1111/codi.14762. Epub 2019 Aug 13. PMID 31309661
- [Background] Wildgaard K, Petersen RH, Hansen HJ, Moller-Sorensen H, Ringsted TK, Kehlet H. Multimodal analgesic treatment in video-assisted thoracic surgery lobectomy using an intraoperative intercostal catheter. Eur J Cardiothorac Surg. 2012 May;41(5):1072-7. doi: 10.1093/ejcts/ezr151. Epub 2011 Dec 21. PMID 22219442
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Marjanski T, Wnuk D, Bosakowski D, Szmuda T, Sawicka W, Rzyman W. Patients who do not reach a distance of 500 m during the 6-min walk test have an increased risk of postoperative complications and prolonged hospital stay after lobectomy. Eur J Cardiothorac Surg. 2015 May;47(5):e213-9. doi: 10.1093/ejcts/ezv049. Epub 2015 Feb 26. PMID 25721817